CLINICAL TRIAL: NCT06678360
Title: Perioperative Impact After Non-cardiac Surgery of Physical Activity on Short- and Long-term Morbidity and Mortality
Brief Title: Perioperative Impact of Physical Activity on Short- and Long-term Morbidity and Mortality
Acronym: PeriopIPA
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, Karolinska Institutet
Other Study IDs: PeriopIPA Karolinska
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: General Surgery; Perioperative Complication; Perioperative Medicine; Physical Inactivity
Keywords: MET-scores; Physical activity; Perioperative mortality
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over 300 million surgeries are performed globally every year. Complications after surgery - infections, cardiovascular conditions, postoperative pulmonary complications and renal impairment - affect survival and quality of life.

Age and co-morbidity are unmodifiable factors, contributing to increased risk of these perioperative complications. However, a modifiable risk factor is physical activity. This study aims to test if self reported physical activity is associated to lower risk of perioperative morbidity and mortality.

DETAILED DESCRIPTION:
Research question: This cohort study investigates if higher levels of self reported physical activity at preoperative assessment is associated to lower risk of complications and lower mortality.

Background: Previous studies of perioperative outcomes in high-income countries indicate that close to 20% had complications within 30 days after surgery, and that around 3% died within 1 yr after surgery. In multiple studies, postoperative complications massively increase risk of 1yr mortality. Whilst perioperative complications are under-reported, they affect length of stay and days at home up to 30 days after surgery (DAH30). DAH30 is a validated, patient-centered outcome measure with prognostic importance due to high sensitivity to changes in surgical risks and the impact of surgical complications.

Data collection: Age, sex, body mass index, co-morbid conditions (using ICD-codes and reported medication) as well as American Society of Anesthesiologists (ASA) physical status classification will be recorded. Exposure: the Metabolic Equivalent of Task Score (MET-score), reported in the electronic health record by the attending anesthesiologist based on patient history in conjunction with the preoperative assessment.

Analysis: The MET-score is the exposure/the dependent variable and the other factors will be used in multivariable analyses.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (equal to or over 18 years) undergoing elective non-cardiac surgery at the two study sites, Karolinska University Hospital Solna and Karolinska University Hospital Huddinge

Exclusion Criteria:

Patients under the age of 18, transplant, day surgery, acute surgery, anesthesia monitoring, brachy therapy and gamma knife interventions. In case of multiple surgeries, only the first will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (equal to or over 18 years) undergoing elective non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 180000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Mortality will be recorded at 30, 60, 90 and 365 days after index surgery
  Death within the time frames described below
DAH30 (Days At Home alive at 30 days) | 30, 90 and 365 days after index surgery,
  DAH30: Patients who are hospitalized for 14 days postoperatively but are alive on day 30 will have DAH30=16. Patients who are hospitalized for five days, then discharged, but return after 10 days for an additional 11-day stay, will have DAH30=14. Anyone who dies within 30 days will have DAH30=0. This outcome measure is validated in several studies and has a significant advantage in that it correlates well with complications, even better than length of stay (LOS).
  We will further record DAH90 and DAH365, calculated as described above.

SECONDARY OUTCOMES:
Length of stay | One year after index surgery
  Number of days in the hospital after index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD, PhD, Principal Investigator — Karolinska Institutet; Arman Valadkhani, MD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Valadkhani A, Sebghati S, Piehl J, Bell M. Impact of Preoperative Functional Capacity on Postoperative Mortality and Morbidity: A Prospective Cohort Study. Anesthesiology. 2026 Mar 1;144(3):525-534. doi: 10.1097/ALN.0000000000005779. Epub 2025 Oct 3. PMID 41043174

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT06678360/Prot_SAP_000.pdf